CLINICAL TRIAL: NCT02112396
Title: Psychosocial Intervention for Relatives of Individuals Suffering From Chronic Alcohol Dependence
Brief Title: Community Reinforcement and Family Training (CRAFT) for Treatment-resistant Individuals With Alcohol Use Disorders
Acronym: CRAFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luebeck (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Hans-Jürgen Rumpf, PD Dr. Hans-Jürgen Rumpf, University of Luebeck
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BMBF-01GX0702; 07-210 (Other: University of Luebeck, Ethics Committee)
Record Dates: First submitted 2014-04-01; First posted 2014-04-14 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Alcohol Dependence; Alcohol Abuse
Keywords: CRAFT; Concerned Significant Others; Contingency management; Reinforcement; Family Intervention
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Intervention (Experimental): Subjects receive 12 sessions of Community Reinforcement and Family Training (CRAFT) immediately after study inclusion
  Interventions: Behavioral: Community Reinforcement and Family Training
- Waiting list group (Other): Waiting list group members receive the Community Reinforcement and Family Training CRAFT intervention after the first follow-up (3 months post study inclusion)
  Interventions: Behavioral: Community Reinforcement and Family Training

INTERVENTIONS:
Behavioral: Community Reinforcement and Family Training — The Intervention is based on the CRAFT literature and includes Building and sustaining motivation of CSOs, functional analysis of problem behaviors, domestic violence precautions (if mandatory), improving communication skills of CSOs, use of negative consequences of drinking behavior, positive reinforcement of clean and sober behavior, strategies to enrich CSOs lives, and strategies for inviting the addicted individual to enter treatment.

SUMMARY:
The present study examines the efficacy of the Community Reinforcement and Family Training (CRAFT) for Concerned Significant Others (CSOs) of individuals with alcohol use disorders (AUDs) using a randomized waiting list (WL) control group. It is hypothesized that after the Intervention group has received CRAFT and prior to the WL- group having received CRAFT, treatment utilization of individuals with AUDs are substantially elevated in the Intervention group.

DETAILED DESCRIPTION:
CRAFT is an evidence-based intervention aiming to promote treatment entry by treatment refusing individuals suffering from addiction by coaching their Concerned Significant others (e.g., family members). The intervention is based on diverse elements such as communication training, contingency management, functional analysis of problem behaviors and strategies to improve the live of CSOs and aims to rearrange contingencies in the natural environment of the drinkers so that clean behavior is reinforced and drinking behavior is effectively discouraged. The intervention was developed for adult CSOs and usually consists of up to 12 weekly face-to-face sessions with a duration of one hour each.

ELIGIBILITY:
Inclusion Criteria:

* CSOs of individuals with an AUD according to the Diagnostic and Statistical Manual (DSM-IV) or the International Classification of Diseases (ICD-10)
* At least 18 years old
* At least 15 hours of contact per week to the addicted individual

Exclusion Criteria:

* History of severe domestic violence
* Current diagnosis of drug- or alcohol dependence of CSO

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2008-08; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Treatment Utilization of relative with AUD | 3 months
  Treatment utilization rates of the individual holding an AUD were assessed at 3-months follow-up

SECONDARY OUTCOMES:
Mental well-being in participating CSO | 3 months
  Mental health status was assessed using the Beck Depression Inventory (BDI) and the Mental Health Inventory (MHI-5)

OTHER OUTCOMES:
Drinking behavior of relative with AUD | 3 months
  Drinking behavior assessed by the AUDIT-C

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Juergen Rumpf, PD Dr., Principal Investigator — University of Luebeck
Locations (1):
- University of Luebeck, Lübeck, Schl.-Holstein, Germany

REFERENCES:
- [Background] Iwen J, Bischof G, Reinhardt S, Grothues J, Hapke U, John U, Freyer-Adam J, Rumpf HJ. The impact of having a loved one with alcohol consumption-related problems on subjective health status and health-risk behaviors in a general hospital sample. Subst Use Misuse. 2010 Dec;45(14):2470-80. doi: 10.3109/10826084.2010.487233. Epub 2010 Jun 10. PMID 20536354